CLINICAL TRIAL: NCT06899269
Title: Proyecto SPAROBOPAN (Registro Nacional De Cirugía Róbotica Pancreática)
Brief Title: SPAROBOPAN Project (Spanish Registry of Robotic Pancreatic Surgery)
Acronym: SPAROBOPAN
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Candido Fernando Alcazar-Lopez, Clinical professor, Hospital General Universitario de Alicante
Other Study IDs: 2024-089
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Robotic Surgical Procedures; Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Duoneopancreatectomy: Resection of the head of the pancreas
  Interventions: Device: robotic resection with Da Vinci Xi
- Distal pancreatectomy: Resection of the body and the tail of the pancreas
  Interventions: Device: robotic resection with Da Vinci Xi
- Total pancreatectomy: Total removal of the pancreas
  Interventions: Device: robotic resection with Da Vinci Xi
- central pancreatectomy: body or neck of the pancreas resection
  Interventions: Device: robotic resection with Da Vinci Xi

INTERVENTIONS:
Device: robotic resection with Da Vinci Xi — robotic resection with Da Vinci Xi

SUMMARY:
Pancreatic robotic surgery (PRS) has moved from an almost testimonial procedure to a moment of expansion that is not yet clearly defined. In the pioneering centres, the results achieved are superior to those of open surgery. At present, it is not known how many centres perform CRP, what type of operations they perform, what percentage of the total number of pancreatic operations CRP represents and what results are obtained. The aim of our project is to establish a national multicentre registry of robotic pancreatic surgery that will allow us to answer all these questions.

Methodology: This is a one-year prospective multicentre registry involving all general and digestive surgery units in Spain that have a DaVinci robotic platform and wish to participate and perform robotic pancreatectomies.

All adult patients undergoing robotic pancreatectomy at participating Spanish centres who meet the inclusion criteria will be included. The registry will be open until 31 March 2026 to include post-operative morbidity and mortality at 90 days. The number of pancreatic surgeries performed in that centre during the same period will be counted to determine the percentage of robotic pancreatic surgery per centre. Intraoperative complications will be measured according to the Satava classification modified by Halls et al. Postoperative complications will be classified according to the Clavien-Dindo classification and the CCI (Comprehensive Complication Index). Pancreatic fistula, postoperative bleeding and delayed gastric emptying were classified according to the ISGPS classification and biliary fistula according to the ISGLS classification.

ELIGIBILITY:
Inclusion Criteria:

* robotic pancreatic resections
* Asa I-III
* Signed informed consent

Exclusion Criteria:

* Less than 18 years old.
* ASA IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who will undergo robotic pancreatic resections
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 90 postoperative days
  Clavien-Dindo Classification
Postoperative complications | 90 postoperative days
  CCI® (Comprehensive Complication Index). 0-100%. 100% represents the death of the patient.
Number of robotic procedures | 1 year
  Number of robotic pancreatic procedures

SECONDARY OUTCOMES:
Experience of each group in robotic pancreatic surgery | 1 year
  Questonnaire answering the number of robotic procedures in 2024.
Textbook outcome | 1 year
  Composite measure: No reintervention, no major complications, no readmission, no pancreatic leak B/C, no mortality and no prolongued hospital stay
Total survival | 3 years
  survival after surgery in months
Disease-free survival | 3 years
  Time from surgery to recurrence

IPD SHARING:
Plan to Share IPD: No
Due to local law with personal data